CLINICAL TRIAL: NCT02056886
Title: Multicentric, National, Prospective, Comparative, Non Randomized Study, Assessing Medico-economic Impact of Three Strategies of Sentinel Lymph Node Analysis in Immediately Operable Breast Cancer
Brief Title: Medico-economic Study of Three Strategies of Sentinel Lymph Node Analysis in Operable Breast Cancer
Acronym: SAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ICO-N-2012-08; 2012-A01504-39 (Other: ANSM)
Record Dates: First submitted 2014-02-05; First posted 2014-02-06 (Estimated); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer; Surgery
Keywords: breast cancer, sentinel lymph node, extemporaneous, OSNA
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- OSNA (Experimental): Intra operative sentinel lymph-node sampling. In this experimental arm, the molecular biology technique is only used through the OSNA technique (One Step Nuclear Acid analysis), and no other classical pathology's diagnosis method such as formalin fixation, then parraffin embedding before slices cutting, hematoxylin-eosin-safran staining or any other immunohistochemical stainings.
  According to the results of the staging procedure, the treatment in this arm is decided in conformity with local and national guidelines in breast cancer treatments.
  SLN detection +/- complementary axillary lymphadenectomy is immediately decided if a tumor invasion is detected within the sentinel LN material.
  Interventions: Procedure: SLN detection +/- complementary axillary lymphadenectomy
- PATHOLOGICAL ANALYSIS (Other): No intra operative examination is performed in this arm, but the final pathological examination:
  In this arm, the classical pathology's diagnosis method is starting with a formalin fixation of suspected invaded lymph-nodes sampling at least 24Hrs; then parraffin embedding before slices cutting; then hematoxylin-eosin-safran staining or any other immunohistochemical stainings.
  According to the results of the staging procedure, the treatment in this arm is decided in conformity with local and national updated guidelines in breast cancer treatments.
  SLN detection +/- complementary axillary lymphadenectomy: is decided in a second surgical step when the pathologic analysis has detected a tumor invasion
  Interventions: Procedure: SLN detection +/- complementary axillary lymphadenectomy
- EXTEMPORANEOUS (Other): "Intra-operative" pathological frozen sections of sentinel LN samples are coloured and examined immediately by the pathologist, allowing an immediate result at the disposal of the surgeon who can decide to complete by an axillary LN dissection or not.
  Then the remaining material will be prepared similarly as in the pathological classical method (Arm B), ie formalin fixation, then parraffin embedding, then slices cutting, then HES staining or ImmunoHistochemistry for a final diagnosis.
  SLN detection +/- complementary axillary lymphadenectomy: is decided immediately when the tumor invasion is detected in the sentinel LN material.
  Interventions: Procedure: SLN detection +/- complementary axillary lymphadenectomy

INTERVENTIONS:
Procedure: SLN detection +/- complementary axillary lymphadenectomy — breast cancer surgery with SLN detection +/- complementary axillary lymphadenectomy Whatever the detection method used in the lab (Arm A: OSNA; Arm B: Pathological Examination; Arm C: Extemporaneous) to assess the positivity of sentinel lymph-node invasion, if negative result (no tumor invasion in the sentinel LN), a complementary lymph-node dissection is not mandatory if positive result (tumor invasion in the sentinel LN), a complementary lymph-node dissection is performed, either immediately (Arm A and C) or in a second surgical procedure (Arm B)
  Other Names: Surgical complementary dissection of axillary lymph-node.

SUMMARY:
Breast carcinoma requires frequently an adjuvant therapy after surgical excision: in this way, one of the major criteria indicating the need of adjuvant chemotherapy is the diagnosis of a metastatic lymph-node invasion, mainly in the axillary field. Axillary surgery is therefore mandatory at the diagnosis of breast carcinoma. For many years, in order to avoid unnecessary complications due to extensive axillary surgery (for instance, arm enlargement by lymphedema), a limited surgery is frequently performed on the first supposed invaded lymph-nodes (LN) called "sentinel" LN technique; if the sentinel LN are not invaded, extensive axillary surgery can be omitted. To decide it during the surgery, removed sentinel LN are cut in 3 to 4 slices which are examined immediately as smears (cytology) or frozen slices (pathology). However, due to hazard in cutting the LN, micro-metastases can be misdiagnosed. That is why a recent molecular biology method has been developed in which the total LN are crushed and blended, then analyzed by OSNA technique (One Step Nuclear Acid analysis) so as to amplify and detect the mRNA coding for cytokeratin-19 protein witnessing the LN metastatic invasion. A standardized automated technique is available with a mean time of 30 to 50 minutes according to the number of analyzed LN.

In 12 international studies (2830 cases) the consistency between OSNA technique and final pathology is of 91 to 98% and the sensitivity seems higher. Less than 5% of all breast carcinomas cells don't express CK-19 protein.

The use of OSNA technique requires a dedicated machine and a skilled pathologist, increasing slightly the operation time; however it allows to avoid the immediate and long-term complications due to the radical LN axillary surgery in case of negativity of the sentinel LN procedure. To date, the three techniques including extemporaneous examinations (OSNA or classical methods) or not (classical pathological analysis) have their own advantages and drawbacks.

"SAGE" study main objective is to compare these three techniques in terms of direct costs and Quality of Life impacts. The superiority of any of these three techniques is not the purpose of SAGE study, but the economic burden of OSNA technique in comparison with the 2 others in the standard setting in France.

Quality of Life and Pain evaluations will be performed immediately after surgery and during the 6 months after.

DETAILED DESCRIPTION:
Today, standard treatment for early Breast carcinoma starts with a surgical step consisting of the tumor resection and sentinel lymph-node (SLN) detection, in order to select patients to be proposed for complementary axillary lymphadenectomy. This requested information may be obtained during the same operation time by intra operative examination, or after surgery with the consequence of a second surgical procedure when lymphadenectomy appears to be indicated. In France, three strategies are currently used for the management of sentinel lymph nodes:

* intra operative pathological frozen section examination followed by final pathological diagnosis,
* intra operative molecular biology using the OSNA technique (One Step Nuclear Acid analysis)
* no intra operative examination, but the final pathological examination. Each of these 3 strategies has advantage and drawbacks and their own cost. With more than 50000 new cases per year in France, Breast carcinoma, thanks to population screening, more and more small tumors are detected where such information about sentinel LN invasion is needed.

Our proposed study is a prospective, cost-effectiveness and comparative non randomised study where three strategies are evaluated in the current practice of the participating teams.

Main Objective :

• to evaluate in each of these 3 strategies for sentinel LN diagnosis, cost-effectiveness and cost-utility (QALY), Quality of Life,…

Secondary Objectives :

* rate of second surgery needed
* rate of mico-metastases or macro-metastases detected to build a decision score,
* follow-up of non re-operated patient despite positive sentinel LN,
* RNA collection from the crushed and blended sentinel LN
* Quality of Life evaluation through the surgical times using QLQ C30 and Br 23 scales.

Medical section :

At pre-operative consultation, patients will be informed to consent participating in our observational study, without any change in their treatment strategy. Inclusion parameters are strictly the same in the three groups.

At the time of surgery, if intra operative examination is planned, patient will be informed that a complete axillary dissection could be indicated.

Included patients will be followed 15 days after surgery and at 3 and 9 months. Then every 6 months during 2 years, then yearly.

Economical section :

Main objective of " SAGE " study is to light up decision maker in striking the balance of each strategy (induced costs and prevented costs) and results in terms of health as expressed by individuals preference depending on different health status, treatment strategies and clinical practice in French centers.

In our study, the medico-economical evaluation on such a quite National scale (17 different centers) takes place in a practice standardization prospect.

General methodology :

In each participating center, one of the 3 strategies for the sentinel LN analysis is currently used (with or without extemporaneous procedure).

Cost-effect evaluation will inventory all undertaken costs in each strategy and all induced positive or negative consequences, both at a qualitative and quantitative level using micro costing and macro costing evaluations. Evaluation of Quality of Life adjusted to health will be included to the cost effect analysis.

In our study, population studied with a localized breast carcinoma, are women aged between 18 and 65 years old and likely to be active : inclusion criteria are strictly the same in the 3 strategies studied.

In our study, we will consider Hospital and Health Insurance point of view. Hospital prospect will identify and value the cost paid by health institution due to the use of any of these 3 techniques.

Insurance Health prospect will value the costs of each treatment strategy including direct costs related to private medical care and not only those to be reimbursed to the hospital.

The study starts at the time of the sentinel LN excision and ends 9 months later, including the post-operative complications and the possible second surgery for axillary LN excision.

At all 920 patients will be included in the 20 participating team.

ELIGIBILITY:
Inclusion Criteria:

1. Infiltrating breast carcinoma histologically proven (lobular, ...)
2. unifocal,
3. T <3 cm (clinical), palpable or non-palpable tumor (smaller than a centimetre allowed),
4. N0 clinical axillary
5. Conservative surgery,
6. GS detection by isotopic or combined method,
7. Age <65 (for more frequent activity), and> 18 years.
8. Social protection
9. Signed Informed consent

Exclusion Criteria:

1. Recurrence of breast carcinoma,
2. History of ipsilateral breast reduction surgery,
3. Radical surgery.
4. History of lumpectomy
5. Neoadjuvant chemotherapy
6. Multi-focality
7. Neoadjuvant hormone therapy
8. < 18 years old
9. Pregnant or nursing patient or of childbearing age without effective contraception,
10. Legal incapacity or limited legal capacity. Medical or psychological conditions not allowing the subject to understand the study and sign the consent.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 858 (Actual)
Dates: Start 2013-10-21 (Actual); Primary Completion 2018-01-02 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Medico-economic study : medical cost between 3 different sentinel lymph node analysis (histological analysis or molecular biology) in the management of patients treated for invasive breast carcinoma. | from surgery to 9 mounths later
  Several phases are differences to compare the costs of three strategies:
  * surgery
  * hospitalization
  * follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Virginie BORDES, MD, Study Director — Institut de Cancérologie de l'Ouest (ICO) - Nantes, France
Locations (17):
- France (17):
  - ICO Paul Papin, Angers
  - Institut Bergonie, Bordeaux
  - Jean Perrin, Clermont-Ferrand
  - Institut du Sein -Clinique Saint-Amé, Lambres-lez-Douai
  - Oscar Lambret, Lille
  - Institut Paoli Calmettes, Marseille
  - HEGP, Paris
  - Institut Curie, Paris
  - CHU, Pierre-Bénite
  - Eugène Marquis, Rennes
  - Henri BECQUEREL, Rouen
  - Institut Curie, Saint-Cloud
  - Clinique Mutualiste, Saint-Etienne
  - Jean-Marc cancérologie CLASSE, Saint-Herblain
  - CHU, Saint-Priest-en-Jarez
  - IUCT-O, Toulouse
  - Institut de Cancérlogie de Lorraine, Vandœuvre-lès-Nancy